CLINICAL TRIAL: NCT04984928
Title: Predicting the Risk of Readmission in Patients With Chronic Heart Failure
Brief Title: Readmission Risk of Patients With Heart Failure.
Acronym: PREDIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0488
Record Dates: First submitted 2021-07-19; First posted 2021-08-02 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Chronic Heart Failure
Keywords: Heart failure; Prediction; Personnalized medicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) is a frequent, serious, and costly chronic disease: it leads to 150,000 hospitalizations each year in France at a cost of 525 million Euros.

It is estimated that 20-40% of these hospitalizations are preventable by known interventions: home telemonitoring, care coordination, therapeutic intensification and therapeutic education. But these interventions only work if patients at high risk of rehospitalization are targeted to individualize management. In these patients, the risk of rehospitalization depends on clinical, biological, socioeconomic, care pathway, and location-related data. Existing predictive tools perform poorly due to three important limitations: non-use of unstructured clinical data, lack of integration of multimodal data, and weakness of the algorithmic approach.

The objective is to design and validate a predictive algorithm for the risk of rehospitalization in heart failure patients, using multiple data sources

ELIGIBILITY:
Inclusion criteria:

* All consecutive adults
* Admitted to Montpellier University Hospital in 2017-2020
* For heart failure

Exclusion criteria:

- age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
30 days all cause readmission rate | day 30
  30 days all cause readmission rate

SECONDARY OUTCOMES:
90 days all cause readmission rate | day 90
  90 days all cause readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Mercier, PU PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC